CLINICAL TRIAL: NCT05107830
Title: Phenotyping of Primary Hyperoxaluria in Children and Adults
Brief Title: Phenotyping of Primary Hyperoxaluria
Acronym: PHENO-HOPLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8071
Record Dates: First submitted 2021-10-13; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Primary Hyperoxaluria
Keywords: Primary hyperoxaluria; Autosomal recessive; Urolithiasis.; Nephrocalcinosis; Renal failure
MeSH Terms: conditions — Hyperoxaluria, Primary; Urolithiasis; Nephrocalcinosis; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
985 / 5000 Résultats de traduction Primary hyperoxaluria is a rare autosomal recessive disease with an estimated prevalence of around 1 to 3 cases per million population. The most frequent attacks are urolithiasis disease and nephrocalcinosis, ultimately leading to end-stage chronic renal failure. The phenotype of this pathology is very heterogeneous, making the diagnosis difficult.

There is currently a significant diagnostic delay. This is potentially due to atypical forms, or to insufficient clinicians' awareness of its research.

However, the early diagnosis of this pathology is essential, since end-stage chronic renal failure can be avoided or at least delayed with early and appropriate management.

The objective of the study is to describe the phenotype of currently diagnosed primary hyperoxaluria, in order to identify the classic presentations but also the characteristics of atypical presentations

ELIGIBILITY:
Inclusion criteria:

* Major or minor subject having undergone genetic research for primary hyperoxaluria between 01/01/2015 and 31/12/2019
* Major subject not having expressed, after information, the reuse of his data for the purposes of this research
* Child and holders of parental authority who have not expressed, after information, the reuse of their data for the purposes of this research

Exclusion criteria:

* Subject (or his parental authority if he is a minor) who has expressed his opposition to participating in the study
* Subject not residing in France
* Subject of foreign nationality
* Subject under tutorship or curatorship
* Subject under safeguard of justice

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Major or minor subject having undergone genetic research for primary hyperoxaluria between 01/01/2015 and 31/12/2019
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Retropsective study of classic presentations of atypical presentations of primitive hyperoxaluria and its characteristics of atypical presentations | Files analysed retrospectively from January 01, 2015 to December 31, 2019 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Néphrologie et Transplantation - Hôpitaux Universitaires de Strasbourg, Strasbourg, France